CLINICAL TRIAL: NCT06599775
Title: Prospective, Single-arm, Multicenter Exploratory Study of Adebrelimab Combined With Chemotherapy, Endoscopic Resection and Sequential Chemoradiotherapy In the Treatment of Inoperable Clinical Staging T1b-2 Esophageal Squamous Cell Carcinoma
Brief Title: Study of Adebrelimab With Chemotherapy, Endoscopy and Sequential Chemoradiotherapy In Inoperable Esophageal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-EC-II-018
Record Dates: First submitted 2024-07-26; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Resectable Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Albumin-Bound Paclitaxel; Carboplatin; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab and chemotherapy combined with endoscopic resection and simultaneous chemoradiotherapy (Experimental): Adebelizumab, an innovative PD-L1 inhibitor, combined with chemotherapy followed by endoscopic resection and subsequent concurrent chemoradiotherapy
  Interventions: Drug: Adebrelimab injection; Drug: Albumin-Bound Paclitaxel; Drug: Carboplatin injection

INTERVENTIONS:
Drug: Adebrelimab injection — Experimental group：Adebrelimab is an innovative PD-L1 inhibitor, monotherapy can improve pathological complete response rates with tolerable safety
  Other Names: SHR-1316
Drug: Albumin-Bound Paclitaxel — Experimental group：combined with Adebrelimab（PD-L1 inhibitor）,and carboplatin followed by endoscopic resection and subsequent simultaneous radiotherapy combined with albumin-bound paclitaxel and carboplatin
  Other Names: Albumin-Bound Paclitaxel injection
Drug: Carboplatin injection — Experimental group：combined with Adebrelimab（PD-L1 inhibitor），and albumin-bound paclitaxel followed by endoscopic resection and subsequent simultaneous radiotherapy combined with albumin-bound paclitaxel and carboplatin
  Other Names: Carboplatin for injection

SUMMARY:
Evaluating the efficacy and safety of PD-L1 (Programmed Death-L1)antibody combined with endoscopy and radiotherapy for inoperable cT1b-2 (clinical stage tumor 1b-2) esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
Previous studies have already confirm immunotherapy combine with chemotherapy can improve pathological complete response rates. Therefore, it is proposed to carry out a study of immuno-combination chemotherapy combined with endoscopic resection and synchronous radiotherapy and chemotherapy in patients with clinical stage cT1-2N0M0 (clinical stage tumor 1b-2 clinical stage nodes 0 stage metastasis 0) to evaluate the efficacy and safety

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent to voluntarily enroll in the study
2. Age 18-75 years
3. Histologically or cytologically confirmed squamous esophageal cancer of the thoracic segment
4. Staging of clinical tumor stage T1b-2N0M0 (according to American Joint Committee on Cancer 8th edition) as judged by the investigator
5. Contraindication to or refusal of oesophagectomy
6. No prior treatment for oesophageal cancer, including radiotherapy, chemotherapy, or surgery
7. Have at least one measurable lesion (RECIST 1.1 criteria)
8. Eastern Cooperative Oncology Group Performance Status score of 0 to 1
9. No contraindication to radiotherapy
10. Adequate organ function on laboratory tests within 14 days prior to the first administration of the drug Blood routine: WBC≥3.0×109/L; ANC≥1.5×109/L; PLT≥100×109/L; HGB≥90 g/L Liver function: AST≤2.5×ULN; ALT≤2.5×ULN; TBIL≤1.5×ULN Renal function: Cr≤1.5×ULN or creatinine clearance rate ≥50 mL/min Coagulation function: International Normalized Ratio ≤1.5, activated partial thromboplastin time ≤1.5×ULN
11. Female subjects of childbearing potential must have a negative blood pregnancy test performed within 72 hours prior to the first dose and not be breastfeeding, and must agree to use effective contraception for the duration of the trial and for 2 months after the last administration of adebrelimab or 6 months after the last administration of chemotherapeutic agent, whichever is longer; for female subjects whose partner is a female of childbearing potential Male subjects should be surgically sterilised or agree to use effective contraception for the duration of the trial and for 2 months after the last administration of adebrelimab or 3 months after the last administration of chemotherapeutic agent, whichever is longer; sperm donation is not permitted during the study.

Exclusion Criteria:

1. Criteria related to treatment history:

   Any treatment for oesophageal cancer, including surgery, radiotherapy, chemotherapy or other antineoplastic agents Ongoing treatment with immunosuppressive drugs, or systemic hormonal drugs for immunosuppression (doses >10 mg/day prednisone or equivalent) within 2 weeks prior to the first use of study drug; inhaled or topical steroids and adrenal glands at doses >10 mg/day prednisone or equivalent are permitted in the absence of active autoimmune disease Corticosteroid replacement Received live attenuated vaccine within 4 weeks prior to first use of study drug Major surgery or severe trauma within 4 weeks prior to first use of study drug.
2. Tumour-related criteria Patients with non-squamous oesophageal cancer Staging not consistent with clinical tumor stage T1b~2N0M0 Other malignancies diagnosed within 5 years prior to first use of study drug, except cured carcinoma in situ of the uterine cervix, basal or squamous cell skin cancers, limited prostate cancer treated with radical surgery, and ductal carcinoma in situ treated with radical surgery

Other criteria:

Presence of any active autoimmune disease or history of autoimmune disease (the following, but not limited to: autoimmune hepatitis, interstitial pneumonitis, uveitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or asthma that has been in complete remission in childhood and does not require any intervention in adulthood are eligible for inclusion; (Subjects with asthma requiring medical intervention with bronchodilators are not eligible for inclusion)

Have a clinical cardiac condition or disease that is not well controlled, such as:

1. New York Heart Association class 2 or higher heart failure;
2. unstable angina pectoris;
3. myocardial infarction within 1 year;
4. clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention Pregnant or breastfeeding women.

   4. Laboratory Tests: Subjects serologically positive for HIV Active hepatitis B (HbsAg positive and hepatitis B virus DNA ≥2000 IU/ml or copy number ≥104/ml) or active hepatitis C (HCV antibody positive and HCV-RNA positive with concomitant need for antiviral therapy) Active tuberculosis.

   5. Presence of allergies and adverse drug events: Presence of allergy or hypersensitivity to monoclonal antibodies Presence of allergic reaction to albumin-bound paclitaxel, carboplatin

   6. Diseases or laboratory abnormalities that, in the opinion of the investigator, may affect the results of the study or are not in the interest of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response of primary lesion | 14 days after endoscopic resection
  defined as the proportion of subjects with no residual tumor in the primary tumor site and histologically negative lymph nodes

SECONDARY OUTCOMES:
Major pathological response | 14 days after endoscopic resection
  defined as the percentage of subjects with <10% residual tumor in the primary tumor site
Overall Survival | From date of signed informed consent until the date of death from any cause, whichever came first, assessed up to 100 months
  Overall Survival
Recurrence free survival | From the time of complete response to the date of recurrence，assessed up to 100 months
  Recurrence free survival
Incidence of Adverse events | through study completion, assessed up to 50 months
  Incidence of Adverse events
Patients' quality of life | through study completion, assessed up to 50 months
  Assessment of patients' quality of life by means of quality of life score questionnaires, such as EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30)